CLINICAL TRIAL: NCT03182751
Title: Does Early Administration of Tranexamic Acid Reduce Blood Loss and Perioperative Transfusion Requirement in Low Energy Hip Fracture Patients?
Brief Title: Does Early Administration of Tranexamic Acid Reduce Blood Loss and Perioperative Transfusion Requirement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brandon James Yuan, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-004988
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Hip Fractures; Intertrochanteric Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into one of two study groups: TXA administration (treatment) or placebo (control). In order to ensure balance on the subject demographics between the two study groups, the subjects will be stratified on gender, age group (<75 vs. ≥75) and body mass index (<30 vs. ≥30). Within each stratum, subjects will be assigned to either the treatment group or control group using an electronic dynamic allocation program housed in a computer application developed by personnel in the Division of Biomedical Statistics and Informatics.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Using dynamic allocation will ensure that the study subjects will remain balanced on the stratification factors and the treatment group assignment throughout the entire subject accrual phase. This system will be utilized by Central pharmacy personnel to generate the treatment group assignments. Medications will then be delivered from the Central Pharmacy to the emergency department in packaging that does not delineate whether it contains placebo or tranexamic acid. Thus, the patient, treating surgeon, emergency department physician, residents, hospitalist group, anesthesiologist, and data collectors will remain blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid Arm (TXA) (Active Comparator): Subjects will be treated with early administration of TXA in the Emergency Department
  Interventions: Drug: Tranexamic Acid (TXA)
- Control Arm (Placebo Comparator): Subjects will be treated with a placebo in the Emergency Department
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — Intravenously via bolus dose of 1g over ten minutes and an additional 1g over the subsequent 8 hours
  Other Names: Cyklokapron
  Arms: Tranexamic Acid Arm (TXA)
Drug: Placebo — Looks exactly like the study drug, but it contains no active ingredient
  Arms: Control Arm

SUMMARY:
Intertrochanteric hip fractures typically result in blood loss from the fracture and require surgery that can cause further blood loss. This study is being done to look at a medication called tranexamic acid which may reduce blood loss and the need for blood transfusions associated with surgery.

DETAILED DESCRIPTION:
The use of TXA in orthopedic trauma patients is an area of current research interest. A 2010 prospective randomized, controlled trial of perioperative TXA demonstrated reduction in transfusion requirements for intertrochanteric hip fractures treated with short, cephalomedullary nails. This was clinically, though not statistically, significant. Investigators recently conducted a randomized, controlled trial at this institution to evaluated the use of TXA in patients with femoral neck fractures treated with hemiarthroplasty or total hip arthroplasty and found clinically, albeit not statistically, significant reduction in transfusion requirement (accepted for publication). Perhaps tempering the effect seen with perioperative administration of TXA is the blood loss that occurs prior to surgery, the so-called "hidden" blood loss that can be as substantial as 1/3 of total blood loss from a hip fracture. This raises the question whether administration of tranexamic acid at the time of initial presentation after fracture could improve the perioperative care of these patients by decreasing the proportion of patients requiring transfusion and decreasing total blood loss.

ELIGIBILITY:
Inclusion Criteria:

* AO/OTA fracture classification 31A
* Surgically treated with sliding hip screw or cephalomedullary nail (short or long)
* Low energy, isolated injury

Exclusion Criteria:

* Intracapsular hip fractures: AO/OTA fracture classification 31B-C
* Polytrauma patients
* Creatinine clearance less than 30 mL/min
* History of unprovoked VTE and/or recurrent VTE
* Known history of Factor V Leiden, protein C/S deficiency, prothrombin gene mutation, anti-thrombin deficiency, anti-phospholipid antibody syndrome, lupus anticoagulant
* Pregnancy or breastfeeding (pregnancy tests will be performed on all patients of child-bearing potential)
* History of CVA, MI, or VTE within the previous 30 days
* Coronary stent placement within the previous 6 months
* Disseminated intravascular coagulation
* Intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Yuan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers that are outside of the primary listed researchers within the primary institution where the investigation is being performed. While we intend the share the overall results of the study through peer review, we do not have our institution's IRB approval to share individual participant data outside of the institution.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm
Started | 64 | 64
Completed | 64 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.1 (13.5) | 79.69 (12.7) | 79.39 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 19 | 19 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 64 | 64 | 128

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Transfused at Least 1 Unit of Packed Red Blood Cells
Description: Transfusion will be considered for all patients with hemoglobin values of less than 8 g/dL with persistent symptoms or history of significant cardiac disease that may render the patient less able to compensate for significant anemia. Blood transfusion will be considered in all patients with hemoglobin less than 7 g/dL, regardless of symptoms.
Time Frame: Length of hospitalization (approximately 3 to 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm
Number analyzed (Participants) | 64 | 64
Participants | 17 | 19

2. Secondary Outcome: Number of Units of Packed Red Blood Cells Transfused
Description: Number of units of packed red blood cells transfused per patient
Time Frame: Length of hospitalization (approximately 3 to 5 days)
Measure: Mean (Standard Deviation); unit: units of packed red blood cells
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm
Number analyzed (Participants) | 17 | 19
units of packed red blood cells | 1.9 (1.9) | 2.3 (1.7)

3. Secondary Outcome: Calculated Blood Loss
Description: Total blood loss per patient measured in milliliters (mL)
Time Frame: Length of hospitalization (approximately 3 to 5 days)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm
Number analyzed (Participants) | 64 | 64
mL | 1600 (1200) | 2000 (1400)

4. Secondary Outcome: Number of Subjects to Experience Symptomatic Venous Thromboembolism (VTE)
Description: Number of subjects to experience symptomatic Venous Thromboembolism (VTE)
Time Frame: Within 6 months of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm
Number analyzed (Participants) | 64 | 64
Participants | 3 | 1

5. Secondary Outcome: Wound Complications
Description: Number of subjects diagnosed with a wound complication
Time Frame: Within 6 months of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm
Number analyzed (Participants) | 64 | 64
Participants | 4 | 1

6. Secondary Outcome: (Myocardial Infarction) MI Diagnosed
Description: Number of subjects diagnosed with a myocardial infarction
Time Frame: Within 6 months of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm
Number analyzed (Participants) | 64 | 64
Participants | 0 | 2

7. Secondary Outcome: Cerebrovascular Accident (CVA) Diagnosed
Description: Number of subjects diagnosed with a cerebrovascular accident
Time Frame: Within 6 months of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm
Number analyzed (Participants) | 64 | 64
Participants | 0 | 3

8. Secondary Outcome: All-cause Mortality
Description: Number of subject deaths
Time Frame: At 6 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm
Number analyzed (Participants) | 64 | 64
Participants | 7 | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 6 months on all participants.
Arm/Group | Tranexamic Acid Arm (TXA) | Control Arm
All-Cause Mortality (participants affected / at risk) | 7/64 | 6/64
Serious Adverse Events (participants affected / at risk) | 8/64 | 7/64
Other Adverse Events (participants affected / at risk) | 0/64 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid Arm (TXA) (N=64) | Control Arm (N=64)
Deep Vein Thrombosis (DVT) (Vascular disorders) | 3 (3) | 1 (1)
Pulmonary Embolism (PE) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Wound Complication (Surgical and medical procedures) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT03182751/Prot_SAP_000.pdf